CLINICAL TRIAL: NCT00087737
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled, Parallel-Group, Flexible-Dose Study of DVS-233 SR and Venlafaxine ER in Adult Outpatients With Major Depressive Disorder
Brief Title: Study Evaluating DVS-233 SR and Venlafaxine ER in Adult Outpatients With Major Depressive Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 3151A1-317
Record Dates: First submitted 2004-07-13; First posted 2004-07-16 (Estimated); Last update posted 2009-08-19 (Estimated); Status verified 2009-08

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major

INTERVENTIONS:
Drug: DVS-233 SR
Drug: Venlafaxine ER

SUMMARY:
To compare the antidepressant efficacy and safety of DVS-233 SR versus placebo in adult outpatients with MDD.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients.
* Sexually active individuals participating in the study must use a medically acceptable form of contraception during the study and for at least 15 days after the last dose of test article
* Subjects must have a primary diagnosis of major depressive disorder

Exclusion Criteria:

* Treatment with DVS-233 SR at any time in the past
* Treatment with venlafaxine (immediate release [IR] or ER) within 90 days of study day 1
* Known hypersensitivity to venlafaxine (IR or ER)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 369 (Actual)
Dates: Primary Completion 2005-05 (Actual); Study Completion 2005-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, MD, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer